CLINICAL TRIAL: NCT04205786
Title: A Randomized Study of Oral Vitamin B12 for the Treatment of Aromatase Inhibitors (AI)-Associated Musculoskeletal Symptoms (AIMSS) in Women With Early Stage Breast Cancer
Brief Title: Vitamin B12 for Aromatase Inhibitors Associated Musculoskeletal Symptoms in Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics requirements, research cancelled
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5119
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: HR-positive Breast Cancer
MeSH Terms: interventions — Vitamin B 12; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial. Participants will be randomly assigned 1:1 to treatment or control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard of Care (Active Comparator): Day 0:
  * Baseline questionnaires: FACT-ES, BPI-SF, Assessment of AI Adherence, Demographics, CRF, and Supplemental Agents Reporting Form
  * Blood collection
  * Continue Usual Care
  Day 45:
  * Repeat of baseline questionnaires with addition of vitamin B12 supplements form and investigational agent accountability record
  * Blood collection
  * Continue Usual Care
  Day 90:
  -Repeat of day 45
  Interventions: Other: Blood collection; Other: Brief Pain Inventory - Short Form survey; Other: FACT-ES Trial Outcome Index (Version 4); Other: Questionnaire to Assess Adherence to Aromatase Inhibitors; Other: Demographics Questionnaire
- Study Medication Group (B12) (Experimental): Day 0:
  * Baseline questionnaires: FACT-ES, BPI-SF, Assessment of AI Adherence, Demographics, CRF, and Supplemental Agents Reporting Form
  * Blood collection
  * Oral intake of Vitamin B12 Daily in the morning
  Day 45
  * Repeat of baseline questionnaires with addition of investigational agent accountability record
  * Blood collection
  * Oral intake of Vitamin B12 Daily in the morning
  Day 90:
  -Repeat of day 45 without additional study drug intake.
  Interventions: Dietary Supplement: Vitamin B12; Other: Blood collection; Other: Brief Pain Inventory - Short Form survey; Other: FACT-ES Trial Outcome Index (Version 4); Other: Questionnaire to Assess Adherence to Aromatase Inhibitors; Other: Demographics Questionnaire

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — Vitamin B12, orally, 2500 mcg, daily, for 90 days
  Arms: Study Medication Group (B12)
Other: Blood collection — Blood collection for laboratory testing will occur within 10 days of signing the consent form, on day 45 +/- 10 days, and on day 90 +/- 10 days. It will include:
  1. Serum B12 levels
  2. CRP
  3. Homocysteine level
  4. MMA
Other: Brief Pain Inventory - Short Form survey — Brief Pain Inventory - Short Form survey
Other: FACT-ES Trial Outcome Index (Version 4) — FACT-ES Trial Outcome Index (Version 4)
Other: Questionnaire to Assess Adherence to Aromatase Inhibitors — Questionnaire to Assess Adherence to Aromatase Inhibitors
Other: Demographics Questionnaire — Demographics Questionnaire

SUMMARY:
Treatment of hormone receptor (HR)-positive breast cancer with Aromatase Inhibitors (AIs) can lead to associated musculoskeletal pain and may cause patients to discontinue important treatment.

This is a randomized controlled trial assessing the affect of Vitamin B12 on AI-associated joint pain and other outcomes. Participants will be randomly assigned 1:1 to treatment or control arm.

The primary objective of this study is:

-To assess whether daily oral Vitamin B12 decreases average joint pain in women with AI-Associated Musculoskeletal Symptoms

Secondary objectives include:

* To investigate whether daily vitamin B12 improves functional quality of life
* To explore the impact of treatment on serum inflammatory cytokine levels (C- reactive protein) between baseline and various points in treatment.

DETAILED DESCRIPTION:
According to the American Cancer Society, there were more than 250,000 new breast cancer cases in 2017. Incidence of breast cancer increases with age, with more than 75% of patients being postmenopausal at the time of diagnosis. In addition, hormone receptors (HR) are over expressed in the majority of breast cancer tumors in postmenopausal women.

Two classes of anti-endocrine therapies are used for treatment of HR-positive breast cancer: tamoxifen and the AIs, which can only be used to treat postmenopausal women because they are ineffective in women with functional ovaries. Joint pain is a significant AI-associated toxicity, affecting as many as 50% of patients. No factors associated with breast cancer treatment (such as chemotherapy) or co-morbid conditions (such as diabetes or body mass index) have been clearly shown to be predictive of the development of joint pain. The cause of AI-associated musculoskeletal symptoms remains elusive but some think it is associated with the direct effects of estrogen deprivation on bone, neurohormonal changes which result in change in pain sensitivity, and immune system changes that alter the circulating or local inflammatory cytokine concentrations.

Some studies report more than 20% of patients are no longer taking their AI chemotherapy regimen because of AI-associated joint pain. As many as 40,000 women are affected by this toxicity in the United States annually and up to 20,000 women discontinue AI therapy because of intolerable joint pain and muscle aches. The current treatment for AI associated musculoskeletal symptoms is limited to oral pain medications and exercise, but, neither intervention has optimal effects, and the long term use of oral pain medication is problematic. Improvement in the treatment of AI associated musculoskeletal symptoms is needed to improve compliance with therapy, and thereby lead to improved breast cancer outcomes and survivorship.

The study team conducted a pilot study (Campbell et al. Breast J, 2018) which suggested that vitamin B12 reduces pain and improves quality of life for participants taking aromatase inhibitors (AIs) who experienced AI-related musculoskeletal symptoms. This study aims to confirm these results in a phase III randomized prospective trial. If confirmed, Vitamin B12 would become a safe and cost-effective option for the treatment of AI-related musculoskeletal symptoms, leading to improved cancer outcomes and survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed estrogen receptor (ER) and/or progesterone receptor (PgR) positive invasive carcinoma of the breast (Stage I-III) with no evidence of metastatic disease (M0).
* Subjects must have completed mastectomy or breast sparing surgery, and must have recovered from all side effects of the surgery. Patients should have recovered from all Grade 2 or higher side effects of chemotherapy and/or radiation therapy with the exception of alopecia and peripheral neuropathy. Concurrent bisphosphonate and trastuzumab therapies are allowed
* Patients must have aromatase inhibitor (AI) associated musculoskeletal symptoms that began or increased after starting AI therapy. New musculoskeletal pain must not be due specifically to fracture or traumatic injury
* Subjects must currently be taking one of the following aromatase inhibitor (AI) doses for at least 14 days prior to registration and plan to continue for at least an additional 180 days after registration:

  * Anastrozole (Arimidex) 1 mg daily OR
  * Letrozole (Femara) 2.5 mg daily OR
  * Exemestane (Aromasin) 25 mg daily
* Patients must be post-menopausal, as defined by at least one of the following:

  --≥ 12 months since their last menstrual period OR
  * Prior bilateral oophorectomy OR
  * Previous hysterectomy with one or both ovaries left in place (or previous hysterectomy in which documentation of bilateral oophorectomy is unavailable) AND (unless ≥ 60 years of age) FSH values consistent with the institutional normal values for the post-menopausal state.
* Performance status: Patients must have ECOG performance status of 0-2 as assessed by MD or RN
* Patients must have no known allergy or hypersensitivity to vitamin B12
* Must have completed the Brief Pain Inventory Short Form (BPI-SF) within 7 days of enrollment (after signing consent, but prior to starting treatment) and have an "average pain" score of at least 24.
* Patients must not have any contraindicated concurrent illnesses including:

  * History of alcohol or other substance abuse or dependence within 365 days prior to enrollment.
  * Chronic liver disease.
  * End stage renal disease.
* Patients who are receiving treatment with narcotics, tramadol, gabapentin, and/or pregabalin must have been taking a stable dose for at least 30 days prior to registration.
* Patients must be able to complete study questionnaires in English.
* Patients who are currently taking vitamin B12 or a multivitamin containing vitamin B12 will be able to participate in the study after having stopped taking the vitamin B12 or the multivitamin containing the B12 for two weeks before day 1 of treatment.
* Patients must be willing to submit blood samples for laboratory testing [to test for Serum Vitamin B12, CRP, homocysteine level, complete blood count (CBC), potassium, and MMA]. Baseline samples must be obtained prior to beginning protocol treatment.
* All patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vitamin B12 or other agents used in this study.
* Subjects with uncontrolled intercurrent illness including, but not limited to chronic liver disease, end stage renal disease, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in average joint pain according to the Brief Pain Inventory - Short Form (BPI- SF) | At baseline, day 45 (+/- 10 days), and at day 90 (+/- 10 days)
  Change in average joint pain according to the Brief Pain Inventory - Short Form (BPI- SF) average pain score. This item has a scale of 0 to 10 with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine"

SECONDARY OUTCOMES:
Change in worst joint pain according to the BPI-SF | At day 90 (+/- 10 days)
  Change in worst joint pain according to the BPI-SF worst (maximum) pain score. This item has a scale of 0 to 10 with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine".
Quality of life (QOL) as measured by Functional Assessment of Cancer Therapy-Endocrine Scale (FACT-ES) | At baseline, day 45 (+/- 10 days), and at day 90 (+/- 10 days)
  Quality of life (QOL) as measured by Functional Assessment of Cancer Therapy-Endocrine Scale (FACT-ES) a 5-point scale (0-4) with 0 being better, 4 being worse.

OTHER OUTCOMES:
Serum inflammatory cytokine levels (C- reactive protein) | At baseline, day 45 (+/- 10 days), and at day 90 (+/- 10 days)
  Serum inflammatory cytokine levels (C- reactive protein)

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Manuscripts, presentations, abstracts